CLINICAL TRIAL: NCT06299046
Title: Evaluation of Operative Bleeding After Robot-assisted Radical Prostatectomy
Brief Title: Bleeding After Robot-assisted Radical Prostatectomy: a Respective Study
Acronym: UROBLOOD01
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Elisa De Lorenzis, Principal Investigator, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: 3235
Record Dates: First submitted 2024-02-28; First posted 2024-03-07 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer; Bleeding; Prostate Adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: robot-assisted radical prostatectomy — surgical removal of the entire prostate and the seminal vesicles, followed by the vescico-urethral anastomosis to restore the continuity of the lower urinary tract performed using Da Vinci Si and Xi Surgical System (Intuitive Surgical, Sunnyvale, California, USA)

SUMMARY:
Nowadays robot-assisted radical prostatectomy (RARP) has become the standard surgical treatment for localised prostate cancer. The robotic approach has been proven superior to open retropubic prostatectomy (ORP) in terms of surgical-related morbidity: RARP has in fact been associated with significantly lower estimated blood loos (EBL), lower transfusion rate, less length of stay, shorter catheterization time, lower risk of Clavien-Dindo grade II and III complications, lower risk of vesicourethral anastomotic stricture and less post-operative pain. The optimal anatomical visualisation and the extraordinary maneuverability, along with the tamponade effect of the pneumoperitoneum, are surely to be deemed responsible of this statistically significant differences.

However, to this day no study has ever investigated the prognostic significance of haematological parameters in terms of predicting perioperative bleeding risk in patients undergoing RARP.

Therefore, the investigators conducted a retrospective non-interventional cohort study to gather evidence concerning the impact of anemia and thrombocytopenia on bleeding risk following this surgical procedure. Furthermore, the investigators evaluated associations between demographical, pathological and surgical factors and hemorrhagic complications.

The investigators retrospectively evaluated all the patients that underwent robot-assisted radical prostatectomy in our Urology Unit from the 1st of January 2017 to the 31th of December 2020. The investigators collected demographic, clinical and pathological data from the medical records of these patients, with particular attention to other known risk-factors for RARP-associated bleeding (e.g.: volume of the prostate, body mass index, smoking status, nerve sparing technique).

Complications were analyzed according to the Clavien- Dindo classification. Bleeding was assessed by considering both the hemoglobin (Hb) drop after surgery and the fluid intraoperatively collected in the suction canister, with all the due adjustments. Moreover, post-operative haemorrhagic complications were evaluated.

The investigators included patients not younger than 18 years old, of which records of a pre-operative full blood count in the 30 days prior to the surgery along with a full blood count the day after were available.

Criteria for exclusion were a history of congenital coagulopathies and/or congenital thrombocytopenia and patients that underwent salvage radical prostatectomy after radiation therapy.

Statistics: EBL and operative time learning curve is studied. Clinical, pathological, intraoperative risk factors analysis for higher EBL is performed by linear regression modelling. Factors are evaluated independently and jointly. Association between each factor above and post-operative outcomes (i.e. post-op bleeding, need of transfusion and hematuria) is also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients aged 18 years or older undergoing RARP at the Urology Unit between 1 January 2017 and 31 December 2020.
* All patients with a pre-operative complete blood count (CBC) in the last 30 days before surgery and a postoperative first-day CBC will be included.

Exclusion Criteria:

* Patients with congenital coagulation defects or congenital thrombocytopenias
* Patients undergoing salvage radical prostatectomy (post-radiotherapy)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Consecutive patients aged 18 years or older undergoing RARP at the Urology Unit between 1 January 2017 and 31 December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Influence of hemoglobin value on haemorrhagic complications | 4 years
  prevalence of post-operative haemorrhagic complications stratifying by presence/absence of anaemia (evaluated in g/dl)
Influence of hematocrit value on haemorrhagic complications | 4 years
  prevalence of post-operative haemorrhagic complications stratifying by pre-operative hematocrit value expressed in %
Influence of platelet count on haemorrhagic complications | 4 years
  prevalence of post-operative haemorrhagic complications stratifying by presence/absence of thrombocytopenia (evaluated in10^9/L)
Influence of blood group on haemorrhagic complications | 4 years
  prevalence of post-operative haemorrhagic complications stratifying patients by blood group

SECONDARY OUTCOMES:
Identification of possibile demographic and surgical predictive factors of haemorrhagic complications | 4 years
  Evaluation of demographic and surgical predictive factors of post-operative haemorrhagic complications

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided